CLINICAL TRIAL: NCT04456361
Title: A Study of Mesenchymal Stem Cells as a Treatment in Patients With Acute Respiratory Distress Syndrome Caused by COVID-19
Brief Title: Use of Mesenchymal Stem Cells in Acute Respiratory Distress Syndrome Caused by COVID-19
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSC-ARDS-001
Record Dates: First submitted 2020-06-23; First posted 2020-07-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-01

CONDITIONS: ARDS, Human; Covid-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 patients (Experimental): Treatment consistsof Mesenchymal Stem Cells administered as a one-time, single-dose therapy via IV infusion at a dose of 1 X 10 8 cells.
  Interventions: Biological: Mesenchymal Stem Cells derived from Wharton Jelly of Umbilical cords

INTERVENTIONS:
Biological: Mesenchymal Stem Cells derived from Wharton Jelly of Umbilical cords — Mesenchymal Stem Cells as a single-dose therapy via IV infusion at a dose of 1 X 10 8 cells.
  Other Names: UCMSC

SUMMARY:
This is a pilot phase, open label, non-randomized study for the treatment of ARDS in patients infected with COVID-19. Subjects will be enrolled and treated with one dose of mesenchymal stem cells and follow-up will occur 90 days post-treatment.

DETAILED DESCRIPTION:
A Study of Mesenchymal Stem Cells as a treatment in Patients with Acute Respiratory Distress Syndrome caused by COVID-19 is a pilot phase, open label, non-randomized study, with a single study center.

The current pandemic caused by the novel virus SARS-CoV-2 has lead to a health care crisis affecting hospitals, hospital workers and health care structure globally. Many countries are dealing with a disrupted infrastructure in health care and imminent economic downfall to an extent that has not been seen in recent years. COVID-19 has lead to a large number of deaths in several countries, and Mexico has not been an exception. Availability of supplies, hospital space and equipment for mechanical ventilation are running critically low, and it has been a challenge for hospitals coping with severe clinical symptoms in COVID-19. This disease is characterized by pneumonia, fever, cough and occasional diarrhea, and the severity has been largely attributed to the high affinity of the virus to Angiotensin-Converting Enzyme 2 (ACE2) as the main receptor, and the Type II Transmembrane Serine Protease TMPRSS2 as the main host protease that mediates S protein activation on primary target cells in the lung and small intestine.

Many agencies and professional societies are working worldwide in developing treatment guidelines to care for patients with COVID-19, since the present treatments are supportive but not yet curative, therefore these guidelines are based on scientific evidence and expert opinion, the use of an array of drugs approved for other indications, as well as multiple investigational agents that are being studied. Lately, Remdesivir, a novel small-molecule adenine nucleotide analogue antiviral drug that has shown efficacy against Ebola virus in rhesus monkeys has shown improvement in patients with oxygen support. The focus of the research for a cure of COVID-19 has been centered on the individual's response in an immunological context, where an over activation of the immune response can cause a production of a large quantity of inflammatory molecules resulting in a cytokine storm with severe physiological consequences. The cytokine storm induces an increase in inflammatory proteins that results in edema, improper oxygen exchange, acute respiratory distress syndrome (ARDS), other organ damage and secondary infection. In recent studies, mesenchymal stem cells (MSCs) have proven to decrease the hyper inflammatory response in the lungs, leading to a steady recovery in patients with ARDS. The use of umbilical cord mesenchymal stem cells (UC-MSCs) may prove a potential effective measure for the treatment of the cytokine storm induced by COVID-19.

A step forward in a treatment strategy for the novel virus infection in humans would be critical for treating COVID-19 and especially ARDS-induced severe pneumonia, which is currently depleting resources around the world. Because efforts to control lung injury via pharmacological agents have been unsuccessful, mesenchymal stem cell (MSC)-based therapy is being investigated, based on the characteristics of MSCs to self-renew in a limitless manner and their multipotency.

Furthermore, MSC-based therapies have demonstrated in the past of having sufficient promising effects in experimental treatment of ARDS via inhibition of alveolar collapse, collagen accumulation, and cell apoptosis in lung tissue. Recent studies found that administrating allogeneic MSCs in patients with ARDS resulted in no pre-specified adverse events, including hypoxemia, cardiac arrhythmia, and ventricular tachycardia. MSCs are currently attracting interest due to source potential, a high proliferation rate, and a painless procedure that is free of ethical issues. Selection of a starting dose of approximately 100 million cells has been chosen to approximate the standard dosage of cells employed in prior clinical studies. This dosage may be adjusted depending on the data generated during the conduction of the study.

MSCs play a positive role mainly in two ways, namely immunomodulatory effects and differentiation abilities. MSCs can secrete many types of cytokines by paracrine secretion or make direct interactions with immune cells, leading to immunomodulation. The immunomodulatory effects of MSCs are triggered further by the activation of TLR receptor in MSCs, which is stimulated by pathogen-associated molecules such as LPS or double-stranded RNA from virus, like the HCoV-19.

There are many pilot studies conducted with MSC transplantation to explore their therapeutic potential for HCoV-19 infected patients, in many of them the pulmonary function and symptoms of patients were significantly improved days after MSC transplantation. Thus, in this study we intend to prove the intravenous transplantation of MSCs as safe and effective for treatment in patients with COVID-19 pneumonia, especially for patients in severe condition.

Primary Objective: To determine the feasibility and safety of intravenously administered MSCs in patients with Acute Respiratory Distress Syndrome.

Secondary Objectives:

To assess preliminary response in respiratory performance in patients with ARDS.

To assess overall survival of patients. To determine mortality rate at 14 days post treatment. To assess clinical and radiological improvements in patients.

Number of Subjects to be studied: 10

Endpoints

Primary Endpoint:

Evaluate Respiratory distress symptoms based on Berlin definition (RR; Oxygen saturation at rest; Arterial partial pressure of oxygen (PaO2) / Fraction of inspiration O2 (FiO2)).

Determine the degree of ground-glass opacity and pneumonia infiltration in imaging studies (X-ray or CT).

Evaluate clinical improvement based on APACHE II Score. Determine mortality rate at 2 weeks post treatment.

Secondary Endpoints:

Adverse events related to MSC infusion (description, timing, grade, seriousness, and relatedness) Hematological decompensation (based on CBC, SQ and metabolic panels) Objective response rate Progression free survival, overall survival, and best overall response rate Determine if any infusion reactions/toxicity occurs

Clinical and radiological parameters will be assessed at Baseline, 2, 4 and 14 day post-treatment, and there will be a 3 month follow-up by telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to provide informed consent or a legally authorized representative.
* Diagnosis of Acute Respiratory Distress Syndrome according to the Berlin Definition following the failing of prior standard therapy, and other available therapies.

Mild: 200 mm Hg < PaO2/FIO2 ≤ 300 mm Hg with PEEP or CPAP ≥ 5 cm H2Oc Moderate: 100 mm Hg < PaO2/FIO2 ≤ 200 mm Hg with PEEP ≥ 5 cm H2O Severe: PaO2/FIO2 ≤ 100 mm Hg with PEEP ≥ 5 cm H2O

* Diagnostic test positive for SARS-CoV-2
* Age ≥ 18 years
* Any man with a partner of child-bearing potential agrees to use adequate contraception which will include two of the following: hormonal or barrier method of birth control, or abstinence prior to study entry, for the duration of study participation, and for 30 days following completion of therapy.

Exclusion Criteria:

* Current or anticipated use of other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MSC infusion plus any patently atopic patients who have a history of having experienced an episode of allergic anaphylaxis.
* Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease).
* Known diagnosis of human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation | Baseline, and at days 2, 4 and 14 post-treatment
  Number of patients with changes in percentage of resting Oxygen saturation (%O2)

SECONDARY OUTCOMES:
Oxygen pressure in inspiration | Baseline, and at days 2, 4 and 14 post-treatment
  Changes in mmHg of Arterial partial pressure of oxygen / Fraction of inspiration O2 (PaO2/FiO2) in all participants
ground-glass opacity | Baseline, and at day 14 post-treatment
  Changes in percentage of participants with reduction in bilateral ground-glass opacities
Pneumonia infiltration | Baseline, and at day 14 post-treatment
  Changes in percentage of participants with reduction of pneumonia bilateral infiltration
Lactate dehydrogenase | Baseline, and at days 4 and 14 post-treatment
  Number of participants with a reduction in Lactate dehydrogenase (mg/dL)
C-reactive protein | Baseline, and at days 4 and 14 post-treatment
  Number of participants with a reduction in C-reactive protein (mg/dL)
D-dimer | Baseline, and at days 4 and 14 post-treatment
  Number of participants with a reduction in D-dimer (mg/dL)
Ferritine | Baseline, and at days 4 and 14 post-treatment
  Number of participants with a reduction in Ferritine (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Perez, Principal Investigator — Instituto de Medicina Regenerativa; Juan Parcero, Study Chair — Instituto de Medicina Regenerativa
Locations (1):
- Instituto de Medicina Regenerativa, Tijuana, Estado de Baja California, Mexico